CLINICAL TRIAL: NCT05611060
Title: Building Healthy Life Skills for Merced County Navigation Center
Brief Title: Evaluation of the Building Healthy Life Skills Program
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Merced (Other)
Responsible Party: Principal Investigator, Linda Diane Cameron, Professor, University of California, Merced
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cameron2022
Record Dates: First submitted 2022-10-29; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Adverse Childhood Experiences; Housing Problems; Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The study utilizes a pretest-posttest design, with surveys completed at baseline immediately prior to the start of the intervention onset, immediately after completion of the intervention, and at follow-up 3 months after the completion of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Building Healthy Life Skills Program — The intervention provides education and training in the long-term mental and physical health consequences of childhood adversity and emotion regulation skills.

SUMMARY:
The goal of this intervention trial is to learn test whether participation in the Building Health Life Skills Program leads to improvements in psychological well-being and stress management skills for people who are experiencing homelessness and housing insecurity. The main questions it aims to answer are:

* Will participation in the Building Healthy Life Skills Program lead to better skills in managing negative emotions?
* Will participation in the Building Healthy Life Skills Program lead to improvements in psychological well-being, sleep quality, and health-related quality of life?

Participants will be asked to complete three surveys: one prior to the first session of the program, one at the end of the program, and one three months later. The surveys include measures of skills for managing negative emotions, mood states, sleep quality, health-related quality of life, illness experiences, and history of childhood adversity.

DETAILED DESCRIPTION:
Community members who are experiencing homelessness and receiving support services from the Merced County Navigation Center and who have enrolled in the center's Building Healthy Life Skills Program will be invited to participate in this intervention evaluation study. The Building Healthy Life Skills program is a 10-week program designed to provide participants with an understanding of how abuse, neglect and household dysfunctions during childhood affect emotional, social, and cognitive well-being; and to provide training in emotion regulation skills, including adaptive emotional processing and expression, mindfulness, and cognitive reappraisal. The sessions are two hours in duration and conducted in classroom style. Open enrollment will be conducted four times a year, serving approximately 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are receiving support services from the Merced County Navigation Center due their current experiences of housing insecurity or homelessness, and
* have enrolled in the Building Healthy Life Skills program

Exclusion Criteria:

* Individuals under the age of 18 years and those who cannot speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life as assessed by the SF-12, for which scores range from 0 to 100 with higher scores reflecting better quality of life | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Health-related quality of life as assessed by the SF 12
Change in depressive symptoms as assessed by the Center for Epidemiological Studies Depression measure, for which averaged rating scores range from 0 to 3 with higher scores reflecting more depressive symptoms | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Center for Epidemiological Studies Depression measure
Change in stress as assessed by the Perceived Stress Scale, for which averaged rating scores range from 1 to 5 with higher scores reflecting greater stress | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Perceived Stress Scale
Change in rumination as an emotion regulation behavior as assessed by the Rumination and Reflections Questionnaire,for which averaged rating scores range from 1 to t with higher scores reflecting more rumination | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Rumination and Reflections Questionnaire
Change in emotional suppression as assessed by the Cortauld Emotional Control Scale (scores range is 1-4, higher scores reflect higher suppression) and the Emotion Regulation Questionnaire (scores range is 1-5, higher scores reflect higher suppression) | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Cortauld Emotional Control Scale and the Emotion Regulation Questionnaire
Change in mindfulness as an emotional regulation tendency as assessed by the Mindful Awareness Attention Scale, for which averaged rating scores range from 1 to 5 with higher scores reflecting greater mindfulness tendencies | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Mindful Awareness Attention Scale
Change in cognitive reappraisal as an emotion regulation strategy as assessed by the Emotion Regulation Questionnaire, for which averaged rating scores range from 1 to 5 with higher scores reflecting higher use of cognitive reappraisal | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Emotion Regulation Questionnaire
Change in general self-efficacy as assessed by the General Self-Efficacy Survey, for which averaged rating scores range from 1 to 5 with higher scores reflecting higher sense of self-efficacy in managing challenging situations | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the General Self-Efficacy Survey
Change in resilience as assessed by the Ego Resilience 89, for which averaged rating scores range from 1 to 5 with higher scores reflecting higher resilience in managing challenging situations | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Ego Resilience 89
Change in sleep quality as assessed by the Pittsburgh Sleep Quality Inventory, for which averaged rating scores range from 0 to 21 with higher scores reflecting poorer sleep quality | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on the Pittsburgh Sleep Quality Inventory
Change in physical health as assessed by self-reported number of sick days in the past month (ranging from 0 to 31) and a the frequency of 17 symptoms each rated 1 to 5 and higher averaged rating scores reflecting higher symptom loads | Assessed at baseline, immediately following completion of the intervention, and 3 months following intervention completion
  Scores on a symptom checklist and number of sick days

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Merced, Merced, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided on the IPD sharing plan at this point in time.